CLINICAL TRIAL: NCT06694038
Title: Comparative Efficacy and Safety of Needle-Knife Fistulotomy Vs. Standard Cannulation in Primary Biliary Access: a Practical Randomized Controlled Trial
Brief Title: Needle-Knife Fistulotomy Vs. Standard Cannulation Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18D.632
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Biliary Obstruction Due to Common Bile Duct Stone; Malignant Bile Duct Obstruction
Keywords: jaundice; bile duct obstruction; abnormal liver enzymes
MeSH Terms: conditions — Jaundice; Cholestasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Cannulation (Active Comparator): Standard Biliary Cannulation
  Interventions: Procedure: standard biliary cannulation
- NKF Cannulation (Experimental): Biliary Cannulation using NKF technique
  Interventions: Procedure: Needle Knife Fistulotomy

INTERVENTIONS:
Procedure: Needle Knife Fistulotomy — Biliary access using needle knife fistulotomy technique
  Arms: NKF Cannulation
Procedure: standard biliary cannulation — standard biliary cannulation
  Arms: Standard Cannulation

SUMMARY:
Needle-knife fistulotomy (NKF) is traditionally used to achieve biliary access when standard cannulation (SC) techniques are unsuccessful. Based on technical factors and the design of prior studies, the literature suggests NKF should be reserved for expert advanced endoscopists. The aim of this study was to evaluate the efficacy and safety of NKF compared to SC for primary biliary access performed by advanced endoscopists with a range of experience including advanced endoscopy trainees.

ELIGIBILITY:
Inclusion Criteria: older than 18 years of age -

Exclusion Criteria: if unable to provide informed consent, pregnant, hemodynamically unstable, with a prior known history of biliary sphincterotomy or ampullectomy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
post ERCP pancreatitis | within 48 hours of the procedure
  Incidence of post ERCP pancreatitis defined as epigastric abdominal pain with lipase more than three times the upper limit of normal occurring within 48 hours of the procedure

SECONDARY OUTCOMES:
Bleeding | within 48 hours
  Significant bleeding was defined as a need for transfusion and/or need for repeat endoscopy for hemostasis
Perforation | within 48 hours
  Perforation, defined by a full thickness defect either seen during endoscopy or on radiological studies post procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospial, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Patients were not asked to consent for the data to be shared with other institutions